CLINICAL TRIAL: NCT05432219
Title: Endoscopic Transoral Retropterygoid Nasopharyngectomy in Recurrent Nasopharyngeal Carcinoma: a Prospective, Single-arm, Exploratory Trial
Brief Title: A Transoral Retropterygoid Approach to Resect Recurrent Nasopharyngeal Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rNPC-SA-ETORP-V1
Record Dates: First submitted 2022-06-16; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Recurrent Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic Transoral Retropterygoid Nasopharyngectomy (Experimental): a novel endoscopic approach to resect nasopharyngeal carcinoma
  Interventions: Procedure: endoscopic surgery

INTERVENTIONS:
Procedure: endoscopic surgery — endoscopic resection of recurrent nasopharyngeal carcinoma via the transoral retropterygoid nasopharyngectomy approach

SUMMARY:
This is a a prospective, single-arm, and exploratory study of endoscopic resection of recurrent nasopharyngeal carcinoma via transoral retropterygoid approach.

DETAILED DESCRIPTION:
The present study explored a novel transoral retropterygoid approach to resect recurrent nasopharyngeal carcinoma, aiming to investigate the effectiveness of this novel approach in the treatment of recurrent nasopharyngeal carcinoma. The primary end point was the margin-negative (R0) resection rate.

ELIGIBILITY:
Inclusion Criteria:

* Pathology or radiography confirmed recurrent nasopharyngeal carcinoma.
* AJCC rT2-T4 which can be surgically removed.
* No distant metastasis.
* aged 18 or more than 18 years old.
* With or without lymph node metastasis, which can be surgically removed.
* No severe restricted mouth opening, and oral approach eligible.
* Sufficient organ function.
* With signed informed consent.
* ECOG score 0-2, and general physical condition can tolerate general anesthesia surgery.

Exclusion Criteria:

* Primary nasopharyngeal carcinoma
* The patient has surgical contraindications: such as severe cardiopulmonary disease and coagulation dysfunction, etc.
* The patient has any situation that may hinder study compliance or the safety during the study period.
* Suffer from uncontrolled disease which could interfere with treatment.
* Uncontrolled active infection.
* Pregnant or breastfeeding women
* There are some other situations that are not suitable for entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Margin-negative (R0) resection rate | once the pathology results come out, up to 14 days
  The rate of the margin-negative resection of the nasopharyngeal carcinoma

SECONDARY OUTCOMES:
Rate of a complete resection based on imaging findings | within 7 days after surgery
  The rate of a complete resection based on postoperative imaging findings
bleeding volume in surgery | From the beginning to the end of the surgery
  The hemorrhage volume during surgery
Operating time | From the beginning to the end of the surgery
  Duration of operating time
Surgery-associated restricted mouth opening | at 30 days post surgery
  The rate of surgery-associated restricted mouth opening
Disease-free survival (DFS) | From the date of enrollment to relapse or metastasis or death from any cause, up to 2 years
  Duration of the disease-free survival after surgery
local recurrence-free survival (LRFS) | From the date of enrollment to local recurrence or death, up to 2 years
  Duration of the local recurrence-free survival (LRFS) after surgery
quality of life-(EORTC QLQ) -C30 version3.0 using European Organisation for Research and Treatment of Cancer quality of life | From the date of enrollment to the end of study, up to2 years
  using European Organisation for Research and Treatment of Cancer quality of life questionaire（EORTC QLQ) - C30 version3.0. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response leve
quality of life-(EORTC QLQ) -H&N35 | From the date of enrollment to the end of study, up to 2 years.
  using European Organisation for Research and Treatment of Cancer quality of life questionaire（EORTC QLQ）- H&N35，All of the scales and single-item measures range in score from 0 to 100. For all the scales and single-items a high score represents a high level of symptomatology or problems
surgery-associated adverse effect | From the date of surgery to the end of study, up to 2 years.
  Using CTCAE Version5.0 to evaluate related adverse effect Using CTCAE Version5.0 to evaluate related adverse effect Using CTCAE Version5.0 to evaluate related adverse effect Using CTCAE Version 5.0 to evaluate surgery-associated adverse effect

CONTACTS AND LOCATIONS:
Overall Officials: Hongmeng Yu, MD,PhD, Principal Investigator — Eye&ENT Hospital, Fudan University